CLINICAL TRIAL: NCT03066401
Title: Respiratory Variations in Diameters of the Inferior Vena Cava and the Internal Jugular Vein to Assess Blood Withdrawal in Patients With Dysmetabolic Hyperferritinemia
Brief Title: Respiratory Variations for Assessing Blood Withdrawal 2
Acronym: ReVAs2
Status: Terminated | Type: Observational
Why Stopped: insufficient inclusion rate
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2013_37; 2013-A01684-41 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-11-09; First posted 2017-02-28 (Actual); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Dysmetabolic Syndrome; Hyperferritinemia; Obese
Keywords: hyperferritinemia; dysmetabolic hyperferritinemia; obese; blood withdrawal; respiratory variations; inferior vena cava; internal jugular vein; ultrasound; ultrasonography; echography
MeSH Terms: conditions — Hyperferritinemia; Obesity | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- obese patients with dysmetabolic hyperferritinemia: PATIENTS: obese patients with dysmetabolic hyperferritinemia undergoing a therapeutic bleeding.
  INTERVENTIONS: The investigators performed ultrasound measurements (echography) and collected clinical parameters before and after a 300 to 500ml therapeutic bleeding, during a standardized respiratory maneuver.
  Interventions: Procedure: echography

INTERVENTIONS:
Procedure: echography — The inferior vena cava and the internal jugular vein diameters were measured by echography before and after blood withdrawal during a standardized respiratory maneuver

SUMMARY:
OBJECTIVES: To investigate whether respiratory variations of the inferior vena cava (ΔIVC) and internal jugular vein (ΔIJV) diameters during standardized breathing (ΔIVCST and ΔIJVST) increase after a therapeutic bleeding in spontaneously breathing and obese patients with dysmetabolic hyperferricemia.

DESIGN: Prospective, monocentric study in the EFS Nord-de-France blood center.

PATIENTS: Obese patients with dysmetabolic hyperferricemia undergoing a therapeutic bleeding.

INTERVENTIONS: The investigators performed ultrasound measures and collected clinical parameters before and after a therapeutic bleeding, during a standardized respiratory maneuver.

MAIN OUTCOME AND MEASURES: The primary endpoint was the ΔIVCST change induced by a 300 to 500ml therapeutic bleeding. The investigators measured the minimal and maximal IVC and IJV diameters during a standardized respiratory maneuver. ΔIVCST and ΔIJVST were calculated as follows: [(maximal diameter - minimal diameter)/maximal diameter].100.

ELIGIBILITY:
Inclusion Criteria:

* adult patients of > or equal 18 years
* dysmetabolic hyperferritinemia
* undergoing a therapeutic blood withdrawal
* health insured
* obese (body mass index > or equal 30Kg/m²)

Exclusion Criteria:

* pregnancy
* transthoracic echogenicity unsuitable for measuring the inferior vena cava diameters
* clinical signs of active exhalation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients with dysmetabolic hyperferritinemia
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
blood withdrawal-induced changes in the respiratory variations of the inferior vena cava during a standardized respiratory maneuver (ΔIVCST) | during a standardized respiratory maneuver, an average 1 hour maximum
  The primary endpoint was the ΔIVCST change induced by a 300 to 500ml therapeutic bleeding. The investigators measured the minimal and maximal IVC diameters during a standardized ventilation. ΔIVCST was calculated as follows: [(maximal diameter - minimal diameter)/maximal diameter].100.

SECONDARY OUTCOMES:
blood withdrawal-induced changes in the respiratory variations of the internal jugular vein during a standardized respiratory maneuver (ΔIJVST) | during a standardized respiratory maneuver, an average 1 hour maximum
  The primary endpoint was the ΔIJVST change induced by a 300 to 500ml therapeutic bleeding. The investigators measured the minimal and maximal IJV diameters during a standardized ventilation. ΔIJVST was calculated as follows: [(maximal diameter - minimal diameter)/maximal diameter].100.

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Preau, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHRU de Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No